CLINICAL TRIAL: NCT04995601
Title: Wearable Technology to Reduce Risk of DVT and Increase Patient Compliance
Acronym: SBIR2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Recovery Force LLC (Industry)
Collaborators: University of Massachusetts, Amherst (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TP1400-04
Record Dates: First submitted 2021-05-29; First posted 2021-08-09 (Actual); Results first posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2023-04

CONDITIONS: Orthopedic Disorder
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Intervention Model Description: This study will have 2 groups, intervention (RF MAC-group 2) and control (usual care for DVT prevention and mobility-group 1) in postoperative total joint replacement patients at two hospitals.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard of Care (No Intervention): Participants will receive DVT prophylaxis using standard intermittent pneumatic compression during postoperative care after total joint replacement.
- Recovery Force MAC (Experimental): Participants will receive DVT prophylaxis using the RF Health MAC during postoperative care after total joint replacement.
  Interventions: Device: RF Health MAC

INTERVENTIONS:
Device: RF Health MAC — The RF Health MAC is a novel device that is applied to the lower legs of patients that provides intermittent active compressions to the calf muscles which results in increased blood flow in the veins, moving blood towards the direction of the heart and reducing the risk of clot formation.
  Arms: Recovery Force MAC

SUMMARY:
The primary purpose of this study is to conduct a multi-site clinical trial of the Recovery Force Movement and Compressions (RF MAC) System. The study is a randomized comparative study of DVT prophylaxis using either standard IPC (Group 1) or the RF MAC system (Group 2) in 300 patients after TJR surgery at two study sites: Tufts Medical Center (Boston, Massachusetts) and Eskenazi Hospital (Indianapolis, Indiana). This study is funded by a Phase II SBIR awarded to Recovery Force from the National Institutes of Health, National Heart, Lung and Blood Institute (R44-HL132624-02).

DETAILED DESCRIPTION:
DVT is the most feared complication of total joint replacement (TJR), with more than 300,000 total hip and 700,000 total knee replacements performed annually in the U.S. Current recommendations for postoperative DVT prophylaxis after TJR include anti-coagulant medications and/or intermittent pneumatic compression (IPC) of the lower limb for a minimum of 10-14 days. Most current IPC devices are non-mobile, making early postoperative mobility, which is especially important in TJR patients, cumbersome and time-consuming. Upon hospital discharge, most patients go home on pharmacologic DVT prophylaxis. Even when at-home external compression therapy is prescribed (IPC or compression stockings), data suggests compliance rates as low as 10-50%.

Recovery Force (RF) has produced the next generation of mechanical DVT prophylaxis, with a mobile device absent of tubes and pumps, stays in place during ambulation, is lightweight and comfortable for continuous wear, and is designed to improve compliance with recommended use. The hypothesis for Phase II is that IPC using the RF1400 will result in improved compliance, support early mobility and result in significantly higher functional mobility after TJR as compared to standard of care.

The research team will conduct a randomized comparative study of DVT prophylaxis using either standard IPC (Group 1) or the RF1400 (Group 2) in 300 patients after TJR surgery. Dr. Karen Giuliano of the University of Massachusetts Amherst will serve as the overall PI for efforts associated with the study sites. This study will include an inpatient phase and an outpatient phase with patients at two clinical sites: Tufts Medical Center and Indiana University School of Medicine, with each site enrolling 150 patients (75 control/75 experimental).

The overall goal of Phase II is to demonstrate that compliance with perscribed use, comfort, and ease-of-use is significantly higher with the RF1400 than with DVT prophylaxis using either standard IPC (in-hospital) or standard-of-care (at-home) in preparation for full commercialization in the TJR market during Phase III. The DVT therapy market is expected to hit $3.8B by 2021, and the US accounts for over 50% of the global market. With the current risk of bleeding from anticoagulant DVT prophylaxis at 5.6%, the commercial impact of this research is that improved patient compliance with the RF1400 DVT prophylaxis will improve postoperative mobility and provide an effective alternative to anticoagulation.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (age 40-85)
* first elective total hip replacement (THR) or first or second (opposite knee) elective total knee replacement (TKA
* speak English
* expected to have a hospital stay of two days or less
* discharge to home from hospital (not a rehabilitation facility)
* must be able to perform self-care
* BMI between 18 and 39
* calf circumference between 11 and 24.5 inches

Exclusion Criteria:

* partial joint replacement, TJR revisions, emergency surgeries
* calf deformities that would not allow proper fit for external compression device
* non-ambulatory
* clinically malnourished or frail/deconditioned
* vulnerable patients (pregnant women, prisoners, homeless and cognitively impaired)
* do not speak English

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care: Participants received DVT prophylaxis using standard intermittent pneumatic compression during postoperative care after total joint replacement.
- Recovery Force MAC: Participants received DVT prophylaxis using the RF Health MAC during postoperative care after total joint replacement.
  RF Health MAC: The RF Health MAC is a novel device that is applied to the lower legs of patients that provides intermittent active compressions to the calf muscles which results in increased blood flow in the veins, moving blood towards the direction of the heart and reducing the risk of clot formation.
Period: Overall Study
Arm/Group | Standard of Care | Recovery Force MAC
Started | 49 | 57
Completed | 49 | 57
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: We used the same analysis population that was described in our research.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Recovery Force MAC | Total
Number analyzed (Participants) | 49 | 57 | 106
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 29 | 59
  >=65 years | 19 | 28 | 47
Age, Continuous [Mean (Full Range); unit: years] | 63.6 [40 to 76] | 64.4 [40 to 82] | 64.0 [40 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 29 | 53
  Male | 25 | 28 | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 49 | 57 | 106
Region of Enrollment [Number; unit: participants]
  United States | 49 | 57 | 106

OUTCOME MEASURES:

1. Primary Outcome: Compliance to Prescribed Use
Description: Compare patient compliance (percentage of prescribed use/24hr) between the standard of care sequential compression device and the Recovery Force Mobility and Compression (MAC) system in a group of total joint replacement patients.
Time Frame: day 1 postoperative joint replacement
Population: Percent Compliance for Day 1 postop
Measure: Mean (Standard Deviation); unit: percentage of prescribed use/24hr
Arm/Group | Standard of Care | Recovery Force MAC
Number analyzed (Participants) | 26 | 48
percentage of prescribed use/24hr | 67.7 (40.1) | 83.3 (25.8)

2. Primary Outcome: Patient-reported Comfort
Description: Compare patient-reported comfort (patient reported outcomes in the hospital-standard of care vs RF MAC-for overall comfort, where higher score is better device performance (5-pt Likert Scale; 1=Strongly disagree, 2=Disagree, 3=Neutral, 4=Agree, 5=Strongly Agree) between the standard of care sequential compression device and the Recovery Force Mobility and Compression (MAC) system in a group of total joint replacement patients.
Time Frame: at the end of 14-day data collection period
Population: Patient reported outcomes in the hospital (Standard of care vs RF MAC) for overall comfort, where higher score is better device performance (5-pt Likert Scale; 1=Strongly disagree, 2=Disagree, 3=Neutral, 4=Agree, 5=Strongly Agree).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care | Recovery Force MAC
Number analyzed (Participants) | 36 | 44
units on a scale | 3.1 (0.5) | 3.5 (0.3)

3. Primary Outcome: Patient-reported Ease-of-use
Description: Compare patient-reported ease-of-use (using the System Usability Scale, with a range of 0-21, where higher score =higher ease of use) between the standard of care sequential compression device and the Recovery Force Mobility and Compression (MAC) system in a group of total joint replacement patients.
Time Frame: at the end of 14-day data collection period
Population: Patient reported ease-of-use (using the System Usability Scale, with a range of 0-21, where higher score =higher ease of use) between the standard of care sequential compression device and the Recovery Force Mobility and Compression (MAC) system in a group of total joint replacement patients.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care | Recovery Force MAC
Number analyzed (Participants) | 36 | 44
units on a scale | 2.6 (0.4) | 2.3 (0.3)

ADVERSE EVENTS:
Time Frame: Adverse events reports were collected through study completion (14 days).
Description: Used standard definitions
Arm/Group | Standard of Care | Recovery Force MAC
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/57
Other Adverse Events (participants affected / at risk) | 0/49 | 0/57

LIMITATIONS AND CAVEATS:
Due to COVID and one of the sites losing their most high volume orthopedic surgeon, this trial was significantly under-enrolled and underpowered

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-30): https://cdn.clinicaltrials.gov/large-docs/01/NCT04995601/Prot_SAP_000.pdf